CLINICAL TRIAL: NCT01049711
Title: Cost-Utility Analysis of Erythropoietin for Anemia Treatmentin Thai End-Stage Renal Disease Patients With Hemodialysis
Brief Title: Cost Utility Analysis of Erythropoietin for Anemia Treatment in Hemodialysis Patients
Acronym: CUAEPO
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: CUAEPO
Record Dates: First submitted 2010-01-11; First posted 2010-01-14 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Renal Failure
Keywords: erythropoietin; hemodialysis; cost utility; incremental cost-effectiveness ratio; Quality adjusted life year; quality of life
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Erythropoietin

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- erythropoietin
  Interventions: Drug: erythropoietin

INTERVENTIONS:
Drug: erythropoietin

SUMMARY:
To study the cost utility analysis of Erythropoietin (EPO) for maintaining the different hemoglobin (Hb) target levels in anemic hemodialysis patient in routine clinical practice.

DETAILED DESCRIPTION:
In Thailand, the studies that were conducted to find the most useful target Hb have not included the cost effectiveness and/or cost utility analyses. The level at which quality of life is maximized and risk is minimized would be the optimal target. Dialysis patients carry higher risk of death than general population. Anemia is the common complication found in dialysis patients that could lead to mortality. Risk of anemia is occurred in HD patients more than CAPD patients because blood loss is less marked and residual renal function maybe better preserved in patients who receive peritoneal dialysis.Although EPO has been included in the National List of Essential Drugs (NLED) for the treatment of anemia caused by end stage renal disease for maintaining the target hemoglobin but the cost of EPO is so expensive. Cost utility analysis is economic technique for assessing the efficiency of healthcare intervention measuring combined outcomes as the effectiveness, i.e., survival and quality of life in combination as quality adjusted life years (QALYs).This study is a benefit measure at the care giving level by using as a part of planning patient management program and at the policy level for decision making.

ELIGIBILITY:
Inclusion Criteria:

* Patients use EPO at least 6 months with titration of EPO therapy is permitted

Exclusion Criteria:

* Patients under 18 years old.
* Patients who have blood transfusion for anemic treatment within 6 months before EPO treatment and before the study starts
* Patients who change the modality of dialysis
* Patients who switch to other anemia treatment method between the study
* Patients who cannot answer the questionnaire and are not willing to participate in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HD patients use EPO at least 6 months with titration of EPO therapy is permitted
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2009-11; Primary Completion 2010-02 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The utility scores of hemodialysis (HD) patients who use EPO to maintain the Hb target level. | 1 year
Cost of HD patients who use EPO to maintain the Hb target level. | 1 year

SECONDARY OUTCOMES:
The incremental cost-effectiveness ratio (calculated as the ratio between the incremental differences in costs and QALYs associated with 2 alternative treatments) of EPO at the different Hb target levels in HD patients in routine clinical practice. | lifetime horizon (Economic evaluation term)

CONTACTS AND LOCATIONS:
Overall Officials: Tanita Thaweethamcharoen, Ph.D, Principal Investigator — Faculty of Medicine, Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok, Thailand